CLINICAL TRIAL: NCT00751335
Title: Prospective, Randomized, Double-blind Cross-over Study Comparing ThermoSmart® to Conventional Heated Humidity in Patients Suing Continuous Positive Airway Pressure
Brief Title: ThermoSmart® Versus Conventional Humidification in Continuous Positive Airway Pressure (CPAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Suburban Lung Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FPHC SLA 2008
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Humidification; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP with ThermoSmart, then CPAP without ThermoSmart (Experimental): CPAP with ThermoSmart is the application of CPAP with heated humidification and a heated breathing tube.
  CPAP without ThermSmart is the application of CPAP with heated humidification without a heated breathing tube.
  Interventions: Device: CPAP with ThermoSmart, then CPAP without ThermoSmart
- CPAP without ThermoSmart, then CPAP with ThermoSmart (Experimental): CPAP with ThermoSmart is the application of CPAP with heated humidification and a heated breathing tube.
  CPAP without ThermSmart is the application of CPAP with heated humidification without a heated breathing tube.
  Interventions: Device: CPAP without ThermoSmart, then CPAP with ThermoSmart

INTERVENTIONS:
Device: CPAP with ThermoSmart, then CPAP without ThermoSmart — CPAP with ThermoSmart is the application of CPAP with heated humidification and a heated breathing tube.
  CPAP without ThermSmart is the application of CPAP with heated humidification without a heated breathing tube.
  Other Names: ThermoSmart
  Arms: CPAP with ThermoSmart, then CPAP without ThermoSmart
Device: CPAP without ThermoSmart, then CPAP with ThermoSmart — CPAP with ThermoSmart is the application of CPAP with heated humidification and a heated breathing tube.
  CPAP without ThermSmart is the application of CPAP with heated humidification without a heated breathing tube.
  Other Names: ThermoSmart
  Arms: CPAP without ThermoSmart, then CPAP with ThermoSmart

SUMMARY:
That ThermoSMart humidification will result in greater compliance (mask on time, objective and subjective sleep quality than conventional humidification.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Previous diagnosis of OSA permitted, but patient must be novel to CPAP and no previous surgical intervention for OSA or treatment with an oral appliance.
3. AHI ≥ 15 OR AHI ≥ 5 + ESS ≥ 10 OR ESS ≥ 10 + a medical co-morbidity
4. Patient willing to give informed consent and follow study protocol.

Exclusion Criteria:

1. Wake resting SpO2 < 90%
2. Patient requires BiLevel PAP or supplemental oxygen
3. The patient is medically unstable (e.g. respiratory or cardiac failure)
4. Patient unwilling to give informed consent or follow study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A Massie, PhD, Principal Investigator — Suburban Lung Asssociates
Locations (1):
- Suburban Lung Associates, Chicago, Illinois, United States

REFERENCES:
- See also: Fisher & Paykel Healthcare — http://fphcare.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All data from this trial has been lost This includes all case report forms and consent forms and therefore, there are no results to report as no data exists
Period: Overall Study
Arm/Group | CPAP With ThermoSmart, Then CPAP Without ThermoSmart | CPAP Without ThermoSmart, Then CPAP With ThermoSmart
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All data from this trial has been lost. This includes all case report forms and consent forms and therefore, there are no results to report as no data exists.
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP With ThermoSmart, Then CPAP Without ThermoSmart | CPAP Without ThermoSmart, Then CPAP With ThermoSmart | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: CPAP Compliance
Time Frame: 1, 4 & 8 weeks
Population: All data from this trial has been lost This includes all case report forms and consent forms and therefore, there are no results to report as no data exists
Arm/Group | CPAP With ThermoSmart, Then CPAP Without ThermoSmart | CPAP Without ThermoSmart, Then CPAP With ThermoSmart
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Subjective & Objective Sleep Parameters
Time Frame: 1, 4 & 8 weeks
Population: as for baseline characteristics
Arm/Group | CPAP With ThermoSmart, Then CPAP Without ThermoSmart | CPAP Without ThermoSmart, Then CPAP With ThermoSmart
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All data for this trial has been lost. All case report forms and consent forms were lost and therefore, there are no results to report as no data exists.
Arm/Group | CPAP With ThermoSmart, Then CPAP Without ThermoSmart | CPAP Without ThermoSmart, Then CPAP With ThermoSmart
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No